CLINICAL TRIAL: NCT02142413
Title: HEart and BRain Interfaces in Acute Ischemic Stroke (HEBRAS) - A Prospective Oberservational Cohort Study
Brief Title: HEart and BRain Interfaces in Acute Ischemic Stroke
Acronym: HEBRAS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other)
Responsible Party: Principal Investigator, Karl Georg Haeusler, Prof., Charite University, Berlin, Germany
Other Study IDs: EA2/033/14
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Stroke; Atrial fibrillation; Holter ECG; cardiac MRI
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers indicating myocardial damage (cardiac Troponin T), autonomic function (Norepinephrine), prediction of atrial fibrillation (BNP).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Ischemic Stroke: Patients older than 18 years with an acute ischemic stroke (according to WHO criteria), stroke onset within 2 days, language: German, MRI compatibility, admission to the stroke unit at the Charité, Campus Benjamin Franklin.

SUMMARY:
The primary aim of this prospective observational study is to investigate whether an enhanced diagnostic MRI work-up (including cardiac MRI, angiography of the aortic arch and the brain-supplying arteries) combined with an in-hospital Holter-ECG of up to 5 days duration leads to a significant increase in relevant pathologic findings with respect to stroke aetiology as compared to the findings obtained by a routine diagnostic work-up (including stroke unit monitoring, 24h-Holter-ECG, echocardiography, Doppler-ultrasound of the brain-supplying arteries) in patients with acute ischemic stroke and no atrial fibrillation according to past medical history or baseline ECG. A better understanding of the stroke aetiology may improve secondary stroke prevention and long term outcome.

DETAILED DESCRIPTION:
Variations and delays in the diagnostic procedures during hospitalization after acute ischemic stroke are still common, and at the same time, stroke aetiology remains cryptogenic in about 20-25% of stroke unit patients. Recent studies have shown that (a) cardiac MRI is now able to detect cardiac sources of embolism (thrombi and aortic plaques) with equal sensitivity as compared to echocardiography, and (b) prolonged ECG monitoring up to several days/weeks/years can significantly increase the detection rate of atrial fibrillation. These developments might allow a faster and more effective diagnostic work-up in patients with acute ischemic stroke compared to standard diagnostic procedures including doppler-ultrasound of the extracranial brain-supplying arteries, echocardiography, 24-h-Holter ECG and stroke unit monitoring. This prospective observational trial therefore aims to assess the detection rate of pathologic findings relevant to stroke aetiology as obtained by an enhanced MRI set-up (including cardiac MRI, MR-angiography of the brain-supplying arteries) and a prolonged Holter-ECG (of up to 5 days after the stroke) in comparison to findings obtained by routine diagnostic procedures after acute stroke.

Moreover, cumulating evidence implies that acute ischemic stroke can lead to cardiac damage. Since the underlying pathophysiological mechanisms are still poorly understood, the HEBRAS study attempts to tackle the relationship between stroke localization (e.g. insular involvement), observed cardiac damage (as indicated by troponin elevation) and activation of autonomic nervous system (as indicated by impairment of heart rate variability and elevated urinary norepinephrine levels), respectively.

Finally, to clarify the prognostic impact of stroke-induced autonomic dysfunction, heart rate variability will be analysed with respect to functional outcome, mortality, recurrent stroke and myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent by the patient
* Acute ischemic stroke, as confirmed by cerebral MRI or CT
* Admission to the stroke unit of the Department of Neurology, Charité, Campus Benjamin Franklin

Exclusion Criteria:

* Atrial fibrillation known by past medical history or documented by routine electrocardiogram (ECG) on hospital admission
* Participation in an interventional clinical trial
* Pre-stroke life expectancy <1 year
* Mechanic heart valve, cardiac pacemaker or other contraindications to undergo MRI
* History of adverse response to MRI contrast agents
* Known Liver disease prior to stroke
* Mild to severe renal dysfunction (creatinine > 1.3 mg/dl (females); creatinine > 1,7 mg/dl (males))
* Severe congestive heart failure (NYHA III or IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the specialized stroke unit at the Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin (CBF), due to an acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Stroke aetiology | From admission to the stroke unit to hospital discharge, or up to 5 days during hospital stay
  Detection rate of pathologic findings relevant to stroke aetiology (i.e. atrial fibrillation, cardiac thrombi, severe carotid stenosis, aortic plaque > 4mm) in patients with acute ischemic stroke obtained by enhanced diagnostic MRI work-up (cardiac MRI, MR-angiography combined with prolonged Holter-ECG of up to 5 days during the in-hospital stay) in comparison to findings obtained by the routine diagnostic work-up at the Department of Neurology; Charité, Campus Benjamin Franklin (consisting of stroke unit monitoring, echocardiography, ultrasound of the brain-supplying arteries, and 24-hour Holter-ECG).

SECONDARY OUTCOMES:
Atrial fibrillation | up to 5 days after hospital discharge
  Rate of first detected paroxysmal atrial fibrillation by prolonged Holter-ECG monitoring (up to 5 days) after hospital discharge.
Stroke localization and cardiac dysfunction | From admission to the stroke unit to hospital discharge, or up to 5 days during hospital stay
  Association of stroke localization (e.g. insular cortex involvement) to autonomic changes (as indicated by elevated urinary norepinephrine levels and heart rate variability) or cardiac dysfunction (as indicated by troponin T serum levels), respectively.
Outcome | day 90 and day 365 after stroke onset
  Association of heart rate variability to poor functional outcome (mRS>2) and mortality at day 90, as well as to the combined endpoint of recurrent ischemic stroke and myocardial infarction or death at day 365.

CONTACTS AND LOCATIONS:
Overall Officials: Karl G Häusler, MD; FESC, Principal Investigator — Charite University, Berlin, Germany; Christian H Nolte, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité, University Medicine Berlin, Berlin, Germany

REFERENCES:
- [Derived] Hellwig S, Krause T, Scheitz JF, Herm J, Grittner U, Jauert N, Fiebach JB, Kasner M, Doehner W, Endres M, Wachter R, Elgeti T, Nolte CH, Haeusler KG. Enhanced diagnostic workup increases pathological findings in patients with acute ischaemic stroke: results of the prospective HEBRAS study. Stroke Vasc Neurol. 2024 Apr 30;9(2):145-152. doi: 10.1136/svn-2022-002179. PMID 37353342
- [Derived] von Rennenberg R, Herm J, Krause T, Hellwig S, Stengl H, Scheitz JF, Elgeti T, Nagel SN, Endres M, Haeusler KG, Nolte CH. Elevation of cardiac biomarkers in stroke is associated with pathological findings on cardiac MRI-results of the HEart and BRain interfaces in Acute Stroke study. Int J Stroke. 2023 Feb;18(2):180-186. doi: 10.1177/17474930221095698. Epub 2022 May 11. PMID 35403503
- [Derived] Haeusler KG, Grittner U, Fiebach JB, Endres M, Krause T, Nolte CH. HEart and BRain interfaces in Acute ischemic Stroke (HEBRAS)--rationale and design of a prospective oberservational cohort study. BMC Neurol. 2015 Oct 22;15:213. doi: 10.1186/s12883-015-0458-2. PMID 26490042